CLINICAL TRIAL: NCT01332253
Title: A Multi-Center, Randomized, Double-Blind, Placebo-Controlled, Single Dose Trial of the Safety and Efficacy of Intravenous Ibuprofen for Treatment of Pain in Pediatric Patients Undergoing Tonsillectomy
Brief Title: Safety and Efficacy of Intravenous Ibuprofen for Treatment of Pain in Pediatric Patients Undergoing Tonsillectomy
Status: Completed | Phase: Phase 3 | Type: Interventional
Sponsor: Cumberland Pharmaceuticals (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Treatment
Other Study IDs: CPI-CL-014
Record Dates: First submitted 2011-04-07; First posted 2011-04-11 (Estimated); Results first posted 2016-11-03 (Estimated); Last update posted 2016-11-03 (Estimated); Status verified 2016-09

CONDITIONS: Tonsillectomy
Keywords: Tonsillectomy, Pediatric
MeSH Terms: interventions — Saline Solution

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: Yes

ARMS (2):
- Intravenous Ibuprofen (Experimental)
  Interventions: Drug: Intravenous ibuprofen
- Normal Saline (Placebo Comparator)
  Interventions: Other: Normal Saline

INTERVENTIONS:
Drug: Intravenous ibuprofen — Participants will receive a single 10mg/kg dose of intravenous ibuprofen diluted in normal saline at the induction of anesthesia.
  Arms: Intravenous Ibuprofen
Other: Normal Saline — Participants will receive a comparable weight based volume of normal saline as a placebo comparator at the induction of anesthesia.
  Arms: Normal Saline

SUMMARY:
The hypothesis is that a single, pre-operative dose of intravenous ibuprofen will significantly reduce post-operative fentanyl use compared to placebo.

ELIGIBILITY:
Inclusion Criteria:

1. Patients between 6 and 17 years of age scheduled to undergo tonsillectomy.

Exclusion Criteria:

1. Have inadequate intravenous access
2. Patients with significant cognitive impairment
3. Active, clinically significant asthma
4. History of allergy or hypersensitivity to any component of intravenous ibuprofen, NSAIDs, aspirin (or related products), cyclooxygenase-2 inhibitors, or fentanyl.
5. Have a history of congenital bleeding diathesis (e.g. hemophilia) or any active clinically significant bleeding
6. Any child with obstructive sleep apnea, defined as an Apnea-Hypopnea Index of greater than or equal to 5.0
7. Have taken investigational drugs within 30 days before clinical trial material administration.
8. Inability to understand the requirements of the study or be unwilling to provide written informed consent (as evidenced by signature on an informed consent document approved by an Institutional Review Board [IRB]) and agree to abide by the study restrictions. Surrogates will be needed for most patients.
9. Refusal to provide written authorization for use and disclosure of protected health information.
10. Be otherwise unsuitable for the study, in the opinion of the Investigator.

Ages: 6 Years to 17 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child
Enrollment: 161 (Actual)
Dates: Start 2011-07; Primary Completion 2012-07 (Actual); Study Completion 2012-08 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Art P Wheeler, MD, Study Director — Cumberland Pharmaceuticals, Inc.
Locations (6):
- United States (6):
  - Advanced ENT & Allergy, Louisville, Kentucky
  - University Hospital, University of Medicine and Dentistry NJ, Newark, New Jersey
  - Southeastern Clinical Research Associates, Charlotte, North Carolina
  - Children's Hospital of Pittsburgh, Pittsburgh, Pennsylvania
  - Comprehensive Pain Specialists, Hendersonville, Tennessee
  - Baylor College of Medicine/Texas Children's Hospital, Houston, Texas

RESULTS

PARTICIPANT FLOW:
Period: Overall Study
Arm/Group | Intravenous Ibuprofen | Normal Saline
Started | 82 | 79
Completed | 82 | 79
Not Completed | 0 | 0

BASELINE CHARACTERISTICS:
Groups:
- Total: Total of all reporting groups
Arm/Group | Intravenous Ibuprofen | Normal Saline | Total
Number analyzed (Participants) | 82 | 79 | 161
Age, Continuous [Mean (Standard Deviation); unit: years] | 10 (3.4) | 9 (3.0) | 9 (3.2)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 31 | 31 | 62
  Male | 51 | 48 | 99
Ethnicity (NIH/OMB) [Count of Participants; unit: Participants]
  Hispanic or Latino | 14 | 13 | 27
  Not Hispanic or Latino | 68 | 66 | 134
  Unknown or Not Reported | 0 | 0 | 0
Race (NIH/OMB) [Count of Participants; unit: Participants]
  American Indian or Alaska Native | 0 | 0 | 0
  Asian | 3 | 0 | 3
  Native Hawaiian or Other Pacific Islander | 0 | 0 | 0
  Black or African American | 8 | 10 | 18
  White | 69 | 68 | 137
  More than one race | 0 | 0 | 0
  Unknown or Not Reported | 2 | 1 | 3
Region of Enrollment [Number; unit: participants]
  United States | 82 | 79 | 161

OUTCOME MEASURES:

1. Primary Outcome: Number of Doses of Fentanyl Administered in the Postoperative Period Prior to Discharge.
Description: To evaluate the primary objective of reduced fentanyl use in the post-operative period, the number of fentanyl doses (0.5 mcg/kg IV) administered in the post-operative period prior to discharge will be measured.
Time Frame: 4 hours
Measure: Mean (Standard Deviation); unit: fentanyl doses
Arm/Group | Intravenous Ibuprofen | Normal Saline
Number analyzed (Participants) | 82 | 79
fentanyl doses | 1.5 (1.32) | 1.7 (1.12)

2. Secondary Outcome: Postoperative Pain as Measured by the Visual Analog Scale (VAS) 30 Minutes Post-procedure.
Description: The patient's self-reported pain at 30 minutes post-procedure will be measured using a VAS scale. The VAS is a continuous scale made up of a horizontal line, 100 mm in length, anchored by 2 verbal descriptors (No Pain, Worst Possible Pain). The VAS is self-completed by the respondent. The subject is asked to place a line perpendicular to the VAS line at the point that represents their pain intensity. Using a ruler, the score is determined by measuring the distance, in mm, on the 100 mm line between the "No Pain" anchor and the subject's mark. The score would be between 0 and 100. A lower score represents less pain while a higher score represents more pain.
Time Frame: 30 minutes post-procedure
Population: Patient reported pain was evaluated utilizing a visual analog scale (VAS) 30 minutes post-procedure.
Measure: Mean (Standard Deviation); unit: millimeters
Arm/Group | Intravenous Ibuprofen | Normal Saline
Number analyzed (Participants) | 82 | 79
millimeters | 51 (30.9) | 55 (27.4)

3. Secondary Outcome: Postoperative Pain as Measured by the Visual Analog Scale (VAS) 60 Minutes Post-procedure.
Description: To evaluate the secondary objective of pain, the patient's self-reported pain at 60 minutes post-procedure will be measured using a VAS scale. The VAS is a continuous scale made up of a horizontal line, 100 mm in length, anchored by 2 verbal descriptors (No Pain, Worst Possible Pain). The VAS is self-completed by the respondent. The subject is asked to place a line perpendicular to the VAS line at the point that represents their pain intensity. Using a ruler, the score is determined by measuring the distance, in mm, on the 100 mm line between the "No Pain" anchor and the subject's mark. The score would be between 0 and 100. A lower score represents less pain while a higher score represents more pain.
Time Frame: 60 minutes post-procedure
Population: Patient reported pain was evaluated utilizing a visual analog scale (VAS) 60 minutes post-procedure.
Measure: Mean (Standard Deviation); unit: millimeters
Arm/Group | Intravenous Ibuprofen | Normal Saline
Number analyzed (Participants) | 82 | 79
millimeters | 39 (27.4) | 47 (30.8)

4. Secondary Outcome: Postoperative Pain as Measured by the Visual Analog Scale (VAS) 90 Minutes Post-procedure.
Description: o evaluate the secondary objective of pain, the patient's self-reported pain at 90 minutes post-procedure will be measured using a VAS scale. The VAS is a continuous scale made up of a horizontal line, 100 mm in length, anchored by 2 verbal descriptors (No Pain, Worst Possible Pain). The VAS is self-completed by the respondent. The subject is asked to place a line perpendicular to the VAS line at the point that represents their pain intensity. Using a ruler, the score is determined by measuring the distance, in mm, on the 100 mm line between the "No Pain" anchor and the subject's mark. The score would be between 0 and 100. A lower score represents less pain while a higher score represents more pain.
Time Frame: 90 minutes post-procedure
Population: Patient reported pain was evaluated utilizing a visual analog scale (VAS) 90 minutes post-procedure.
Measure: Mean (Standard Deviation); unit: millimeters
Arm/Group | Intravenous Ibuprofen | Normal Saline
Number analyzed (Participants) | 82 | 79
millimeters | 29 (29.3) | 35 (30.8)

5. Secondary Outcome: Postoperative Pain as Measured by the Visual Analog Scale (VAS) 120 Minutes Post-procedure.
Description: To evaluate the secondary objective of pain, the patient's self-reported pain at 120 minutes post-procedure will be measured using a VAS scale. The VAS is a continuous scale made up of a horizontal line, 100 mm in length, anchored by 2 verbal descriptors (No Pain, Worst Possible Pain). The VAS is self-completed by the respondent. The subject is asked to place a line perpendicular to the VAS line at the point that represents their pain intensity. Using a ruler, the score is determined by measuring the distance, in mm, on the 100 mm line between the "No Pain" anchor and the subject's mark. The score would be between 0 and 100. A lower score represents less pain while a higher score represents more pain.
Time Frame: 120 minutes post-procedure
Population: Patient reported pain was evaluated utilizing a visual analog scale (VAS) 120 minutes post-procedure.
Measure: Mean (Standard Deviation); unit: millimeters
Arm/Group | Intravenous Ibuprofen | Normal Saline
Number analyzed (Participants) | 82 | 79
millimeters | 22 (26.2) | 27 (29.3)

6. Secondary Outcome: Time to Discharge Post Procedure.
Description: To evaluate the secondary objective of pain, the time to participant discharge will be measured.
Time Frame: Discharge
Measure: Mean (Standard Error); unit: hours
Arm/Group | Intravenous Ibuprofen | Normal Saline
Number analyzed (Participants) | 82 | 79
hours | 1.9 (0.10) | 1.9 (0.11)

7. Secondary Outcome: Time to Swallow Post Procedure.
Description: Swallowing will be assessed every 15 minutes following arrival to the recovery room; the time to first swallow will be recorded.
Time Frame: every 15 minutes until able to swallow
Measure: Mean (Standard Error); unit: hours
Arm/Group | Intravenous Ibuprofen | Normal Saline
Number analyzed (Participants) | 82 | 79
hours | 0.5 (0.04) | 0.4 (0.03)

8. Secondary Outcome: Parent Satisfaction With Regards to Pain Management Post Procedure.
Description: To evaluate the secondary objective of pain, parental satisfaction during the post-operative period will be measured with regards to pain management. The Parental Satisfaction Survey asked the parent to base their response on their child's management from the time they arrive in the recovery room until they were discharged. Question 1 asked "How satisfied were you with your child's pain management at the time of discharge?"
Time Frame: Discharge
Population: Summary of Parent Satisfaction Post-Procedure with Pain Management at the time of discharge?
Measure: Number; unit: participants
Arm/Group | Intravenous Ibuprofen | Normal Saline
Number analyzed (Participants) | 73 | 65
participants
  Strongly Agree | 58 | 58
  Agree | 11 | 6
  Neutral | 1 | 1
  Disagree | 2 | 0
  Strongly Disagree | 0 | 0
  Survey question not completed | 1 | 0

9. Secondary Outcome: Parent Satisfaction With Regards to Nausea Management Post Procedure.
Description: To evaluate the secondary objective of pain, parental satisfaction during the post-operative period will be measured with regards to nausea management. The Parental Satisfaction Survey asked the parent to base their response on their child's management from the time they arrive in the recovery room until they were discharged. Question 2 asked "How satisfied were you with your child's nausea management during the study?"
Time Frame: Discharge
Population: Summary of Satisfaction Post-Procedure with nausea management during the study
Measure: Number; unit: participants
Arm/Group | Intravenous Ibuprofen | Normal Saline
Number analyzed (Participants) | 73 | 65
participants
  Strongly Agree | 64 | 57
  Agree | 7 | 5
  Neutral | 0 | 2
  Disagree | 0 | 0
  Strongly Disagree | 0 | 0
  Survey question not completed | 2 | 1

10. Secondary Outcome: Parental Satisfaction With Vomiting Control in the Post-Operative Period.
Description: To evaluate the secondary objective of pain, parental satisfaction during the post-operative period will be measured with regards to vomiting control. The Parental Satisfaction Survey asked the parent to base their response on their child's management from the time they arrive in the recovery room until they were discharged. Question 3 asked "How satisfied were you with your child's vomiting management during the study?"
Time Frame: Discharge
Population: Summary of Satisfaction Post-Procedure with Vomiting Control.
Measure: Number; unit: participants
Arm/Group | Intravenous Ibuprofen | Normal Saline
Number analyzed (Participants) | 73 | 65
participants
  Strongly Agree | 66 | 59
  Agree | 3 | 4
  Neutral | 1 | 2
  Disagree | 0 | 0
  Strongly Disagree | 0 | 0
  Survey question not completed | 3 | 0

11. Secondary Outcome: Blood Loss During Surgery
Description: Amount of Blood Lost During Surgery in milliliters
Time Frame: End of Surgery
Population: Blood loss during surgery in milliliters
Measure: Mean (Standard Deviation); unit: milliliters
Arm/Group | Intravenous Ibuprofen | Normal Saline
Number analyzed (Participants) | 82 | 79
milliliters | 15 (29.6) | 16 (39.3)

ADVERSE EVENTS:
Arm/Group | Intravenous Ibuprofen | Normal Saline
Serious Adverse Events (participants affected / at risk) | 1/82 | 0/79
Other Adverse Events (participants affected / at risk) | 7/82 | 10/79
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Intravenous Ibuprofen (N=82) | Normal Saline (N=79)
Tonsillar haemorrhage (Respiratory, thoracic and mediastinal disorders) | 1 (1) | 0 (0)
OTHER ADVERSE EVENTS (reported when occurring in more than 3% of participants in an arm); cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Intravenous Ibuprofen (N=82) | Normal Saline (N=79)
Vomiting (Gastrointestinal disorders) | 3 (3) | 2 (2)
Agitation (Nervous system disorders) | 1 (1) | 3 (3)
Restlessness (Nervous system disorders) | 0 (0) | 2 (2)
Rash Erythematous (Skin and subcutaneous tissue disorders) | 0 (0) | 2 (2)
Infusion Site Pain (Injury, poisoning and procedural complications) | 3 (3) | 0 (0)
Bronchospasm (Immune system disorders) | 0 (0) | 2 (2)

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: No